CLINICAL TRIAL: NCT05125588
Title: Randomized, Single-dose, Crossover, Two-period, Two-sequence, Laboratory-blinded, Comparative Bioavailability Study of Meloxicam 15 mg Tablets in Healthy Volunteers Under Fasting Condition.
Brief Title: Fasting Comparative Bioavailability Study of 2 Meloxicam 15 mg Tablets in Healthy Volunteers Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joint Stock Company "Farmak" (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FM-MEL
Record Dates: First submitted 2021-11-15; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Pharmacokinetics
Keywords: bioequivalence; pharmacokinetics; generic drugs; Meloxicam
MeSH Terms: interventions — Meloxicam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Reumoxicam® 15 mg tablets (PJSC "Farmak", Ukraine)
  Interventions: Drug: Reumoxicam® 15 mg tablets (PJSC "Farmak", Ukraine)
- Treatment B (Active Comparator): Movalis 15 mg tablets ("Boehringer Ingelheim Ellas A.E.", Greece)
  Interventions: Drug: Movalis 15 mg tablets ("Boehringer Ingelheim Ellas A.E.", Greece)

INTERVENTIONS:
Drug: Reumoxicam® 15 mg tablets (PJSC "Farmak", Ukraine) — One tablet was administered orally and swallowed at once, without chewing, by study volunteers, followed by 200 ml of water, under fasting condition (after preliminary nocturnal fasting for 12 hours) in the morning at 8:00 hours on Day I Period I and Period II of the study.
  Other Names: Meloxicam
  Arms: Treatment A
Drug: Movalis 15 mg tablets ("Boehringer Ingelheim Ellas A.E.", Greece) — One tablet was administered orally and swallowed at once, without chewing, by study volunteers, followed by 200 ml of water, under fasting condition (after preliminary nocturnal fasting for 12 hours) in the morning at 8:00 hours on Day I Period I and Period II of the study.
  Other Names: Meloxicam
  Arms: Treatment B

SUMMARY:
The aim of the study was to compare the bioavailability of two formulations of meloxicam given to healthy volunteers and to demonstrate bioequivalence. The test product, Reumoxicam® 15 mg tablets (Farmak PJSC, Ukraine), given in a single dose was compared with a licensed reference product Movalis 15 mg tablets ("Boehringer Ingelheim Ellas A.E.", Greece), in a randomized, laboratory-blind, single dose, two periods, crossover study.

The secondary objective of the trial was to investigate the safety of both preparations on the basis of safety clinical and laboratory examinations (at the beginning and at the end of the trial) and registration of adverse events and/ or adverse drug reactions.

DETAILED DESCRIPTION:
Randomized, single-dose, crossover, two-period, two-sequence, laboratory-blinded, comparative bioavailability study of test medicinal product Reumoxicam® 15 mg tablets (PJSC "Farmak", Ukraine) and reference medicinal product Movalis 15 mg tablets ("Boehringer Ingelheim Ellas A.E.", Greece) in healthy volunteers under fasting condition.

During each period 18 blood samples were taken: before dosing (0) and then at: 0.5; 1; 2; 3; 4; 4.5; 5; 5.5; 6; 7; 8; 10; 12; 24; 36; 48 and 72 hours after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers, men and women aged 18 to 45 years (inclusive);
2. Provided written Informed Consent Form of a Healthy Volunteer for Participation in the Clinical Study before the beginning of any screening procedures;
3. Ability (to the opinion of the investigator) to fulfill all requirements of the Study Protocol, i.e. the volunteer's ability for adequate collaboration;
4. Body mass index is within the limits (> 18,5 kg/m2 and < 30,0 kg/m2);
5. Persons free from any acute and chronic diseases of cardiovascular system, neuroendocrine system, kidneys, liver, gastrointestinal tract, and respiratory system;
6. Results of physical, instrumental, and laboratory examination of volunteers are within the normal limits, or any deviations are classified by the investigator as clinically irrelevant;
7. Chest fluorography or radiography results are within the normal limits (the examination should be carried out no earlier than 9 months before the screening moment), or any deviation is classified by the investigator as clinically irrelevant;
8. Women and men have to use medically confirmed barrier method of contraception during the whole study period;
9. Volunteers have to be non-smokers or smoke up to 10 cigarettes a day inclusive;
10. Volunteers need to undertake to follow all general diet limitations during the whole study period.

Exclusion Criteria:

1. Subjects with evidence or suspicion of any relevant clinical abnormality (as based on medical history, physical examination, vital signs, chest X-ray, and 12-lead ECG)
2. Known hypersensitivity to meloxicam and/or other investigational products ingredients;
3. Compromised allergologic history;
4. Subjects who have developed signs of asthma, nasal polyps, angio-oedema or urticaria following the administration of aspirin or other NSAIDs;
5. Active peptic ulcer, gastrointestinal perforation or bleeding within the last 6 months;
6. Subjects with peripheral oedema;
7. Any previously incurred diseases or surgical interventions which, to the investigator's opinion, may affect pharmacokinetics of the investigational product;
8. Positive result of HIV, syphilis, hepatitis B and C markets test;
9. Positive result of urine test for narcotic substances (amphetamine, metamphetamine, morphine, marijuana, cocaine);
10. Positive result of alcohol vapors test in expired air;
11. Pregnancy (positive result of urine pregnancy test in women) and lactation period;
12. Incurred acute infectious diseases within 28 days before beginning of the study;
13. Use of any medicinal products within 14 days before beginning of the study;
14. Blood donation or blood loss of more than 300 ml in less than 30 days before beginning of the study;
15. Participation in any other clinical study during the last 90 days before beginning of the study;
16. Other reasons which, to the investigator's opinion, make the volunteer's participation in the study undesirable.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01-29 (Actual); Primary Completion 2014-02-26 (Actual); Study Completion 2014-02-26 (Actual)

PRIMARY OUTCOMES:
AUC0-t | up to 72 hours post-administration
  Area under the plasma concentration-time curve from time zero to time t of the last quantifiable concentration
Cmax | up to 72 hours post-administration
  Maximum drug concentration in plasma

SECONDARY OUTCOMES:
AUC0-inf | up to 72 hours post-administration
  Area under the plasma concentration-time curve from time zero to infinity
tmax | up to 72 hours post-administration
  time after administration to reach maximum drug concentration in plasma
t1/2 | up to 72 hours post-administration
  elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Udovytskyi, Study Chair — Joint Stock Company "Farmak"

IPD SHARING:
Plan to Share IPD: No